CLINICAL TRIAL: NCT01313858
Title: Non-Interventional Study Investigating the Use of Golimumab (Simponi®) in Patients With Rheumatoid Arthritis, Psoriatic Arthritis, and Ankylosing Spondylitis
Brief Title: A Study to Investigate the Use of Golimumab (Simponi®) in Participants With Rheumatoid Arthritis, Psoriatic Arthritis and Ankylosing Spondylitis (P06554)
Acronym: GO-NICE
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P06554; MK-8259-005 (Other: Merck)
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Results first posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-09

CONDITIONS: Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylitis, Ankylosing
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylitis, Ankylosing | interventions — golimumab; Methotrexate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Participants with Rheumatoid Arthritis: Simponi®-naïve participants with rheumatoid arthritis given Simponi® 50 mg once a month as a subcutaneous injection. Combination use with methotrexate was recommended.
  Interventions: Drug: Simponi®; Drug: Methotrexate
- Participants with Psoriatic Arthritis: Simponi®-naïve participants with psoriatic arthritis given Simponi® 50 mg once a month as a subcutaneous injection.
  Interventions: Drug: Simponi®
- Participants with Ankylosing Spondylitis: Simponi®-naïve participants with ankylosing spondylitis given Simponi® 50 mg once a month as a subcutaneous injection.
  Interventions: Drug: Simponi®

INTERVENTIONS:
Drug: Simponi®
  Other Names: Golimumab
Drug: Methotrexate — Given concomitantly with Simponi®
  Groups: Participants with Rheumatoid Arthritis

SUMMARY:
This is a study to assess the use of golimumab (Simponi®) in participants with rheumatoid arthritis, psoriatic arthritis, and ankylosing spondylitis. The study objective is to evaluate the clinical safety of golimumab (Simponi®) under real-life, clinical practice conditions as assessed by the incidence and type of (serious) adverse events and changes in clinical status of participants as assessed by clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Has rheumatoid arthritis, psoriatic arthritis, or ankylosing spondylitis and treatment with Simponi® by autoinjector device is to be initiated for the first time

Exclusion Criteria:

* No specific exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in a primary care clinic or office with rheumatoid arthritis, psoriatic arthritis, or ankylosing spondylitis for whom the treatment with Simponi® by autoinjector device is to be initiated for the first time
Sampling Method: Non-Probability Sample
Enrollment: 1613 (Actual)
Dates: Start 2010-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Kruger K, Burmester GR, Wassenberg S, Thomas MH. Golimumab as the First-, Second-, or at Least Third-Line Biologic Agent in Patients with Rheumatoid Arthritis, Psoriatic Arthritis, or Ankylosing Spondylitis: Post Hoc Analysis of a Noninterventional Study in Germany. Rheumatol Ther. 2020 Jun;7(2):371-382. doi: 10.1007/s40744-020-00204-9. Epub 2020 Apr 17. PMID 32303994
- [Derived] Kruger K, Burmester GR, Wassenberg S, Bohl-Buhler M, Thomas MH. Patient-reported outcomes with golimumab in patients with rheumatoid arthritis, psoriatic arthritis, and ankylosing spondylitis: non-interventional study GO-NICE in Germany. Rheumatol Int. 2019 Jan;39(1):131-140. doi: 10.1007/s00296-018-4180-4. Epub 2018 Nov 10. PMID 30415451
- [Derived] Kruger K, Burmester GR, Wassenberg S, Bohl-Buhler M, Thomas MH. Effectiveness and safety of golimumab in patients with rheumatoid arthritis, psoriatic arthritis and ankylosing spondylitis under real-life clinical conditions: non-interventional GO-NICE study in Germany. BMJ Open. 2018 Jun 14;8(6):e021082. doi: 10.1136/bmjopen-2017-021082. PMID 29903793

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis | Participants With Ankylosing Spondylitis
Started | 524 | 546 | 543
Completed | 238 | 276 | 305
Not Completed | 286 | 270 | 238
Not completed — Premature Treatment Termination | 251 | 219 | 191
Not completed — Lost to Follow-up | 35 | 51 | 47

BASELINE CHARACTERISTICS:
Population: The Modified Intention to Treat Population (mITT) population consists of all participants who were treated with Simponi® and have a baseline assessment and at least one additional visit, regardless of any protocol violations during the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis | Participants With Ankylosing Spondylitis | Total
Number analyzed (Participants) | 474 | 501 | 483 | 1458
Age, Continuous [Mean (Standard Deviation); unit: Years] — The mITT population consists of all participants who were treated with Simponi® and have a baseline assessment and at least one additional visit, regardless of any protocol violations during the study.
  Years | 54.9 (13.38) | 50.3 (12.07) | 43.6 (12.29) | 49.6 (13.39)
Sex: Female, Male [Count of Participants; unit: Participants] — The mITT population consists of all participants who were treated with Simponi® and have a baseline assessment and at least one additional visit, regardless of any protocol violations during the study.
  Participants
    Female | 345 | 271 | 162 | 778
    Male | 129 | 230 | 321 | 680

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression (CGI) Disease Status
Description: The CGI is a non-disease-specific evaluation of participants' overall health status assessed on a 10 mm visual analogue scale (VAS) ranging from "0" (free of complaints) to "10" (strong discomfort). The closer the score to 0, the better the health status.
Time Frame: Baseline (BL; Month 0), Month 3, Month 6, Month 9, Month 12, Month 15, Month 18, Month 21, Month 24
Population: The mITT population consists of all participants who were treated with Simponi® and have a baseline assessment and at least one additional visit, regardless of any protocol violations during the study.
Measure: Least Squares Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 474 | 501 | 483
Units on a scale
  BL | 5.7 (2.21) [3.69 to 6.74] | 5.5 (2.17) [2.77 to 6.01] | 5.7 (2.19) [3.69 to 6.74]
  Month 3 | 3.4 (2.27) [4.10 to 7.33] | 3.2 (2.25) [2.71 to 6.08] | 2.9 (2.13) [4.10 to 7.33]
  Month 6 | 3.1 (2.25) [4.13 to 7.58] | 2.8 (2.19) [3.80 to 7.44] | 2.5 (2.09) [4.13 to 7.58]
  Month 9 | 2.7 (1.99) [4.50 to 8.08] | 2.6 (2.07) [4.97 to 8.77] | 2.4 (1.87) [4.50 to 8.08]
  Month 12 | 2.8 (2.11) [6.21 to 9.82] | 2.4 (2.01) [3.98 to 7.89] | 2.3 (1.94) [6.21 to 9.82]
  Month 15 | 2.5 (1.89) | 2.3 (1.96) | 2.2 (1.85)
  Month 18 | 2.4 (1.97) | 2.2 (1.86) | 2.2 (1.91)
  Month 21 | 2.5 (1.99) | 2.1 (1.84) | 2.2 (1.78)
  Month 24 | 2.2 (1.84) | 2.1 (1.95) | 2.1 (2.01)

2. Primary Outcome: Change From Baseline in FFbH (Funktionsfragebogen Hannover) Questionnaire Score
Description: The FFbH is a participant questionnaire assessing disability/functional impairment. Ability to perform 18 activities of daily living are scored on a 3 point scale (2=Yes, 1=Yes but with effort, and 0=No or with assistance) and summed. Remaining functional capacity is calculated as the percent of the maximum number of score points (FFbH[%] = (Attained score*100)/(2*n) where n is the number of completed responses) with range from 0 = total loss of functional capacity to 100 = maximal functional capacity. Increase from baseline in FFbH score signifies improvement. The FFbH is similar to Health Assessment Questionnaire (HAQ) but is more widely used in Germany.
Time Frame: Baseline and Months 3, 6, 9, 12, 15, 18, 21, 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 474 | 501 | 483
Units on a scale
  Month 3 (n=348;361;375) | 5.29 (1.56) [2.23 to 8.34] | 5.82 (1.54) | 8.66 (1.31)
  Month 6 (n=263;310;297) | 5.71 (1.69) [2.40 to 9.30] | 6.31 (1.61) | 10.01 (1.40)
  Month 9 (n=226;265;262) | 5.78 (1.77) | 7.07 (1.69) | 9.67 (1.45)
  Month 12 (n=218;247;247) | 5.70 (1.79) | 7.86 (1.73) | 8.34 (1.48)
  Month 15 (n=188;222;234) | 5.63 (1.89) | 6.64 (1.79) | 9.04 (1.50)
  Month 18 (n=168;211;216) | 6.98 (1.96) | 8.99 (1.82) | 8.79 (1.54)
  Month 21 (n=166;198;200) | 5.43 (1.97) | 9.18 (1.86) | 7.95 (1.59)
  Month 24 (n=167;198;211) | 7.42 (1.97) | 7.71 (1.86) | 9.51 (1.56)
Statistical Analysis 1: Comparison: Participants With Rheumatoid Arthritis; Least squares mean difference from baseline in FFbH at Month 3 (Month 3 minus BL); Test type: Superiority or Other; p = 0.0007, Repeated measures analysis
Statistical Analysis 2: Comparison: Participants With Rheumatoid Arthritis; Least squares mean difference from baseline in FFbH at Month 6 (Month 6 minus BL); Test type: Superiority or Other; p = 0.0007, Repeated measures analysis
Statistical Analysis 3: Comparison: Participants With Rheumatoid Arthritis; Least squares mean difference from baseline in FFbH at Month 9 (Month 9 minus BL); Test type: Superiority or Other; p = 0.0011, Repeated measures analysis
Statistical Analysis 4: Comparison: Participants With Rheumatoid Arthritis; Least squares mean difference from baseline in FFbH at Month 12 (Month 12 minus BL); Test type: Superiority or Other; p = 0.0015, Repeated measures analysis
Statistical Analysis 5: Comparison: Participants With Rheumatoid Arthritis; Least squares mean difference from baseline in FFbH at Month 15 (Month 15 minus BL); Test type: Superiority or Other; p = 0.0029, Repeated measures analysis
Statistical Analysis 6: Comparison: Participants With Rheumatoid Arthritis; Least squares mean difference from baseline in FFbH at Month 18 (Month 18 minus BL); Test type: Superiority or Other; p = 0.0004, Repeated measures analysis
Statistical Analysis 7: Comparison: Participants With Rheumatoid Arthritis; Least squares mean difference from baseline in FFbH at Month 21 (Month 21 minus BL); Test type: Superiority or Other; p = 0.0059, Repeated measures analysis
Statistical Analysis 8: Comparison: Participants With Rheumatoid Arthritis; Least squares mean difference from baseline in FFbH at Month 24 (Month 24 minus BL); Test type: Superiority or Other; p = 0.0002, Repeated measures analysis
Statistical Analysis 9: Comparison: Participants With Psoriatic Arthritis; Least squares mean difference from baseline in FFbH at Month 3 (Month 3 minus BL); Test type: Superiority or Other; p = 0.0002, Repeated measures analysis
Statistical Analysis 10: Comparison: Participants With Psoriatic Arthritis; Least squares mean difference from baseline in FFbH at Month 6 (Month 6 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 11: Comparison: Participants With Psoriatic Arthritis; Least squares mean difference from baseline in FFbH at Month 9 (Month 9 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 12: Comparison: Participants With Psoriatic Arthritis; Least squares mean difference from baseline in FFbH at Month 12 (Month 12 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 13: Comparison: Participants With Psoriatic Arthritis; Least squares mean difference from baseline in FFbH at Month 15 (Month 15 minus BL); Test type: Superiority or Other; p = 0.0002, Repeated measures analysis
Statistical Analysis 14: Comparison: Participants With Psoriatic Arthritis; Least squares mean difference from baseline in FFbH at Month 18 (Month 18 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 15: Comparison: Participants With Psoriatic Arthritis; Least squares mean difference from baseline in FFbH at Month 21 (Month 21 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 16: Comparison: Participants With Psoriatic Arthritis; Least squares mean difference from baseline in FFbH at Month 24 (Month 24 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 17: Comparison: Participants With Ankylosing Spondylitis; Least squares mean difference from baseline in FFbH at Month 3 (Month 3 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 18: Comparison: Participants With Ankylosing Spondylitis; Least squares mean difference from baseline in FFbH at Month 6 (Month 6 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 19: Comparison: Participants With Ankylosing Spondylitis; Least squares mean difference from baseline in FFbH at Month 9 (Month 9 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 20: Comparison: Participants With Ankylosing Spondylitis; Least squares mean difference from baseline in FFbH at Month 12 (Month 12 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 21: Comparison: Participants With Ankylosing Spondylitis; Least squares mean difference from baseline in FFbH at Month 15 (Month 15 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 22: Comparison: Participants With Ankylosing Spondylitis; Least squares mean difference from baseline in FFbH at Month 18 (Month 18 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 23: Comparison: Participants With Ankylosing Spondylitis; Least squares mean difference from baseline in FFbH at Month 21 (Month 21 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 24: Comparison: Participants With Ankylosing Spondylitis; Least squares mean difference from baseline in FFbH at Month 24 (Month 24 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis

3. Primary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score
Description: The FACIT-F scale assesses self-reported fatigue and its impact upon daily activities and function. 13 items consisting of fatigue, weakness, listlessness, tiredness, trouble with starting things, trouble with finishing things, energy, activity, sleep, eating, help doing activities, frustration, and social activities are scored on a scale of 0 (not at all) to 4 (very much), except energy and activity which are reversed scored. Individual item scores are then summed to provide the final FACIT-F score with range from 0 (lowest) to 52 (highest quality of life). Increase from baseline in FACIT-F score signifies improvement.
Time Frame: Baseline and Months 3, 6, 12, 18, 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 474 | 501 | 483
Units on a scale
  Month 3 (n=344;356;368) | 2.85 (0.79) [3.69 to 6.74] | 4.39 (0.83) [2.77 to 6.01] | 5.21 (0.78) [3.69 to 6.74]
  Month 6 (n=264;311;300) | 3.71 (0.85) [4.10 to 7.33] | 4.40 (0.86) [2.71 to 6.08] | 5.71 (0.82) [4.10 to 7.33]
  Month 12 (n=215;242;243) | 4.81 (0.91) [4.13 to 7.58] | 5.62 (0.93) [3.80 to 7.44] | 5.86 (0.88) [4.13 to 7.58]
  Month 18 (n=167;212;216) | 5.05 (0.99) [4.50 to 8.08] | 6.87 (0.97) [4.97 to 8.77] | 6.29 (0.91) [4.50 to 8.08]
  Month 24 (n=162;196;211) | 5.99 (1.00) [6.21 to 9.82] | 5.94 (1.00) [3.98 to 7.89] | 8.01 (0.92) [6.21 to 9.82]
Statistical Analysis 1: Comparison: Participants With Rheumatoid Arthritis; Least squares mean difference from baseline in FACIT-F at Month 3 (Month 3 minus BL); Test type: Superiority or Other; p = 0.0003, Repeated measures analysis
Statistical Analysis 2: Comparison: Participants With Rheumatoid Arthritis; Least squares mean difference from baseline in FACIT-F at Month 6 (Month 6 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 3: Comparison: Participants With Rheumatoid Arthritis; Least squares mean difference from baseline in FACIT-F at Month 12 (Month 12 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 4: Comparison: Participants With Rheumatoid Arthritis; Least squares mean difference from baseline in FACIT-F at Month 18 (Month 18 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 5: Comparison: Participants With Rheumatoid Arthritis; Least squares mean difference from baseline in FACIT-F at Month 24 (Month 24 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 6: Comparison: Participants With Psoriatic Arthritis; Least squares mean difference from baseline in FACIT-F at Month 3 (Month 3 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 7: Comparison: Participants With Psoriatic Arthritis; Least squares mean difference from baseline in FACIT-F at Month 6 (Month 6 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 8: Comparison: Participants With Psoriatic Arthritis; Least squares mean difference from baseline in FACIT-F at Month 12 (Month 12 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 9: Comparison: Participants With Psoriatic Arthritis; Least squares mean difference from baseline in FACIT-F at Month 18 (Month 18 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 10: Comparison: Participants With Psoriatic Arthritis; Least squares mean difference from baseline in FACIT-F at Month 24 (Month 24 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 11: Comparison: Participants With Ankylosing Spondylitis; Least squares mean difference from baseline in FACIT-F at Month 3 (Month 3 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 12: Comparison: Participants With Ankylosing Spondylitis; Least squares mean difference from baseline in FACIT-F at Month 6 (Month 6 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 13: Comparison: Participants With Ankylosing Spondylitis; Least squares mean difference from baseline in FACIT-F at Month 12 (Month 12 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 14: Comparison: Participants With Ankylosing Spondylitis; Least squares mean difference from baseline in FACIT-F at Month 18 (Month 18 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 15: Comparison: Participants With Ankylosing Spondylitis; Least squares mean difference from baseline in FACIT-F at Month 24 (Month 24 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis

4. Primary Outcome: Change From Baseline in EuroQol- 5 Dimension 3 Level Version (EQ-5D-3L) Questionnaire Score
Description: The EQ-5D-3L is a health profile questionnaire that assesses quality of life along 5 dimensions. Participants rate 5 aspects of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) by choosing from 3 answering options (1=no problems; 2=some problems; 3=extreme problems). The summed score ranges from 1-15 with "1" corresponding to no problems and "15" corresponding to severe problems in the 5 dimensions. Decrease from baseline in EQ-5D-3L signifies improvement.
Time Frame: Baseline and Months 6, 12, 18, 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 474 | 501 | 483
Units on a scale
  Month 6 (n=254;302;293) | -0.69 (0.15) [3.69 to 6.74] | -1.07 (0.14) [2.77 to 6.01] | -1.18 (0.14) [3.69 to 6.74]
  Month 12 (n=211;236;242) | -0.97 (0.16) [4.10 to 7.33] | -1.35 (0.15) [2.71 to 6.08] | -1.24 (0.14) [4.10 to 7.33]
  Month 18 (n=161;206;211) | -1.11 (0.17) [4.13 to 7.58] | -1.35 (0.16) [3.80 to 7.44] | -1.25 (0.15) [4.13 to 7.58]
  Month 24 (n=162;191;210) | -1.08 (0.17) [4.50 to 8.08] | -1.29 (0.17) [4.97 to 8.77] | -1.51 (0.15) [4.50 to 8.08]
Statistical Analysis 1: Comparison: Participants With Rheumatoid Arthritis; Least squares mean difference from baseline in EQ-5D-3L at Month 6 (Month 6 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 2: Comparison: Participants With Rheumatoid Arthritis; Least squares mean difference from baseline in EQ-5D-3L at Month 12 (Month 12 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 3: Comparison: Participants With Rheumatoid Arthritis; Least squares mean difference from baseline in EQ-5D-3L at Month 18 (Month 18 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 4: Comparison: Participants With Rheumatoid Arthritis; Least squares mean difference from baseline in EQ-5D-3L at Month 24 (Month 24 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 5: Comparison: Participants With Psoriatic Arthritis; Least squares mean difference from baseline in EQ-5D-3L at Month 6 (Month 6 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 6: Comparison: Participants With Psoriatic Arthritis; Least squares mean difference from baseline in EQ-5D-3L at Month 12 (Month 12 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 7: Comparison: Participants With Psoriatic Arthritis; Least squares mean difference from baseline in EQ-5D-3L at Month 18 (Month 18 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 8: Comparison: Participants With Psoriatic Arthritis; Least squares mean difference from baseline in EQ-5D-3L at Month 24 (Month 24 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 9: Comparison: Participants With Ankylosing Spondylitis; Least squares mean difference from baseline in EQ-5D-3L at Month 6 (Month 6 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 10: Comparison: Participants With Ankylosing Spondylitis; Least squares mean difference from baseline in EQ-5D-3L at Month 12 (Month 12 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 11: Comparison: Participants With Ankylosing Spondylitis; Least squares mean difference from baseline in EQ-5D-3L at Month 18 (Month 18 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis
Statistical Analysis 12: Comparison: Participants With Ankylosing Spondylitis; Least squares mean difference from baseline in EQ-5D-3L at Month 24 (Month 24 minus BL); Test type: Superiority or Other; p < 0.0001, Repeated measures analysis

5. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event
Description: An adverse event is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure.
Time Frame: Up to 24 months
Population: The safety population consists of all participants with at least one injection of Simponi®.
Measure: Number; unit: Participants
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 524 | 546 | 543
Participants | 320 | 309 | 281

6. Primary Outcome: Number of Participants Who Experienced at Least One Serious Adverse Event
Description: A serious adverse event is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure that results in death, life-threatening adverse event, permanent or significant disability / unfitness for work, hospital treatment (i.e., admission to hospital) or prolongation of a patient's length of stay, or congenital deformity or birth defect.
Time Frame: Up to 24 months
Population: The safety population consists of all participants with at least one injection of Simponi®.
Measure: Number; unit: Participants
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 524 | 546 | 543
Participants | 75 | 70 | 59

ADVERSE EVENTS:
Time Frame: Up to 24 months
Description: Adverse events are described for the safety population consisting of all participants with at least one injection of Simponi®. Results are reported for the entire study population, not for the individual reporting groups according to underlying disease indication.
Groups:
- All Participants: Simponi®-naïve participants with rheumatoid arthritis, psoriatic arthritis, or ankylosing spondylitis given Simponi® 50 mg once a month as a subcutaneous injection.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 204/1613
Other Adverse Events (participants affected / at risk) | 315/1613
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=1613)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1)
NORMOCHROMIC NORMOCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 1 (1)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
CARDIOVASCULAR INSUFFICIENCY (Cardiac disorders) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 5 (5)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1)
SINOATRIAL BLOCK (Cardiac disorders) | 1 (1)
TACHYARRHYTHMIA (Cardiac disorders) | 1 (1)
ACUTE VESTIBULAR SYNDROME (Ear and labyrinth disorders) | 1 (1)
EXOSTOSIS OF EXTERNAL EAR CANAL (Ear and labyrinth disorders) | 1 (1)
HYPOACUSIS (Ear and labyrinth disorders) | 1 (1)
EXOPHTHALMOS (Eye disorders) | 1 (1)
EYELID OEDEMA (Eye disorders) | 1 (1)
PAROPHTHALMIA (Eye disorders) | 1 (1)
RETINAL DETACHMENT (Eye disorders) | 1 (1)
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1)
ENTERITIS (Gastrointestinal disorders) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1)
ILEUS (Gastrointestinal disorders) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1)
MELAENA (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
SUBILEUS (Gastrointestinal disorders) | 1 (1)
SWOLLEN TONGUE (Gastrointestinal disorders) | 1 (1)
CHEST DISCOMFORT (General disorders) | 1 (1)
CHILLS (General disorders) | 1 (1)
CONDITION AGGRAVATED (General disorders) | 2 (2)
DEATH (General disorders) | 4 (4)
DRUG INEFFECTIVE (General disorders) | 1 (1)
FACIAL PAIN (General disorders) | 1 (1)
FATIGUE (General disorders) | 1 (1)
MASS (General disorders) | 1 (1)
PAIN (General disorders) | 2 (2)
PYREXIA (General disorders) | 4 (4)
HEPATIC CYST (Hepatobiliary disorders) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 1 (1)
ATYPICAL PNEUMONIA (Infections and infestations) | 1 (1)
BRONCHITIS (Infections and infestations) | 2 (2)
BRONCHOPNEUMONIA (Infections and infestations) | 2 (2)
CELLULITIS (Infections and infestations) | 2 (2)
CHLAMYDIAL INFECTION (Infections and infestations) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 1 (1)
ENCEPHALITIC INFECTION (Infections and infestations) | 1 (1)
ERYSIPELAS (Infections and infestations) | 1 (1)
FEBRILE INFECTION (Infections and infestations) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (1)
KIDNEY INFECTION (Infections and infestations) | 1 (1)
LOBAR PNEUMONIA (Infections and infestations) | 1 (1)
PERITONITIS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 7 (7)
PULMONARY SEPSIS (Infections and infestations) | 1 (1)
PULMONARY TUBERCULOSIS (Infections and infestations) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1)
SALPINGO-OOPHORITIS (Infections and infestations) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
SINOBRONCHITIS (Infections and infestations) | 1 (1)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 4 (4)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 2 (2)
JOINT INJURY (Injury, poisoning and procedural complications) | 1 (1)
LACERATION (Injury, poisoning and procedural complications) | 1 (1)
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
PERIPROSTHETIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1)
SKULL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 1 (1)
ANTI-CYCLIC CITRULLINATED PEPTIDE ANTIBODY POSITIVE (Investigations) | 1 (1)
COLONOSCOPY (Investigations) | 1 (1)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 2 (2)
HAEMOGLOBIN DECREASED (Investigations) | 1 (2)
INVESTIGATION (Investigations) | 1 (1)
PLATELET COUNT INCREASED (Investigations) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1)
ANKYLOSING SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 3 (3)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
ARTHROFIBROSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
FACET JOINT SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1)
HAND DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 4 (4)
JAW CYST (Musculoskeletal and connective tissue disorders) | 1 (1)
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 (1)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 2 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 4 (4)
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 (1)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 2 (3)
VERTEBRAL FORAMINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CHOLESTEATOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
CHRONIC MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
FIBROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
GASTROINTESTINAL STROMAL TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LIP AND/OR ORAL CAVITY CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
PROSTATIC ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
SALIVARY GLAND NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BURNING SENSATION (Nervous system disorders) | 1 (2)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1 (1)
CEREBELLAR INFARCTION (Nervous system disorders) | 3 (3)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 4 (4)
CEREBROVASCULAR DISORDER (Nervous system disorders) | 1 (1)
CUBITAL TUNNEL SYNDROME (Nervous system disorders) | 1 (1)
DEMYELINATION (Nervous system disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 4 (4)
FACIAL PARESIS (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
MONOPARESIS (Nervous system disorders) | 2 (2)
SCIATICA (Nervous system disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 4 (4)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1)
BURNOUT SYNDROME (Psychiatric disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 2 (3)
MAJOR DEPRESSION (Psychiatric disorders) | 1 (1)
CALCULUS URETERIC (Renal and urinary disorders) | 2 (2)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1)
NEUROGENIC BLADDER (Renal and urinary disorders) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 2 (2)
EPIDIDYMITIS (Reproductive system and breast disorders) | 1 (1)
MENORRHAGIA (Reproductive system and breast disorders) | 3 (3)
VAGINAL EROSION (Reproductive system and breast disorders) | 1 (1)
ALVEOLITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 (4)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 2 (3)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 (1)
PSORIASIS (Skin and subcutaneous tissue disorders) | 2 (2)
PUSTULAR PSORIASIS (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 2 (2)
AUTONOMIC GANGLIONECTOMY (Surgical and medical procedures) | 1 (1)
BLADDER OPERATION (Surgical and medical procedures) | 1 (1)
BURSA REMOVAL (Surgical and medical procedures) | 1 (1)
CARDIAC OPERATION (Surgical and medical procedures) | 1 (1)
CHOLECYSTECTOMY (Surgical and medical procedures) | 2 (2)
CHOLESTEATOMA REMOVAL (Surgical and medical procedures) | 1 (1)
DRUG THERAPY CHANGED (Surgical and medical procedures) | 1 (1)
ENDOMETRIAL ABLATION (Surgical and medical procedures) | 1 (1)
FOOT OPERATION (Surgical and medical procedures) | 1 (1)
GALLBLADDER OPERATION (Surgical and medical procedures) | 1 (1)
HIP ARTHROPLASTY (Surgical and medical procedures) | 3 (3)
HOSPITALISATION (Surgical and medical procedures) | 11 (11)
HYSTERECTOMY (Surgical and medical procedures) | 2 (2)
JOINT ARTHROPLASTY (Surgical and medical procedures) | 1 (1)
KNEE ARTHROPLASTY (Surgical and medical procedures) | 5 (5)
KNEE OPERATION (Surgical and medical procedures) | 2 (2)
LAXATIVE SUPPORTIVE CARE (Surgical and medical procedures) | 1 (1)
LIMB OPERATION (Surgical and medical procedures) | 1 (1)
POLYPECTOMY (Surgical and medical procedures) | 1 (2)
PROSTHESIS IMPLANTATION (Surgical and medical procedures) | 1 (1)
RADIOACTIVE IODINE THERAPY (Surgical and medical procedures) | 1 (1)
SHOULDER ARTHROPLASTY (Surgical and medical procedures) | 2 (2)
SHOULDER OPERATION (Surgical and medical procedures) | 1 (1)
SPINAL DECOMPRESSION (Surgical and medical procedures) | 1 (1)
SPINAL FUSION SURGERY (Surgical and medical procedures) | 1 (1)
SPINAL OPERATION (Surgical and medical procedures) | 1 (1)
SYNOVECTOMY (Surgical and medical procedures) | 4 (6)
TENDON SHEATH INCISION (Surgical and medical procedures) | 2 (2)
TENOTOMY (Surgical and medical procedures) | 1 (1)
TOE OPERATION (Surgical and medical procedures) | 1 (1)
VARICOSE VEIN OPERATION (Surgical and medical procedures) | 1 (1)
VASCULAR GRAFT (Surgical and medical procedures) | 2 (2)
WRIST SURGERY (Surgical and medical procedures) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2)
HYPERTENSION (Vascular disorders) | 1 (1)
HYPERTENSIVE CRISIS (Vascular disorders) | 2 (2)
LYMPHOEDEMA (Vascular disorders) | 2 (2)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 (1)
VENOUS INSUFFICIENCY (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=1613)
DRUG INEFFECTIVE (General disorders) | 315 (315)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No